CLINICAL TRIAL: NCT06340360
Title: A Phase 2b, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Rezpegaldesleukin in the Treatment of Severe to Very Severe Alopecia Areata in Adult Patients (Rezolve AA)
Brief Title: A Phase 2b Study to Evaluate Rezpegaldesleukin (Rezpeg) in the Treatment of Severe to Very Severe Alopecia Areata in Adult Patients (Rezolve AA)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-358-06; 2023-509981-39 (EudraCT Number)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 1 of 3 groups (low dose, high dose, or placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Rezpegaldesleukin Low Dose Every 2 weeks
  Interventions: Drug: Rezpegaldesleukin
- High Dose (Experimental): Rezpegaldesleukin High Dose Every 2 weeks
  Interventions: Drug: Rezpegaldesleukin
- Placebo (Placebo Comparator): Placebo Every 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rezpegaldesleukin — Pharmaceutical form: Injection solution Route of administration: subcutaneous
  Other Names: REZPEG; NKTR-358; LY3471851 (formerly)
  Arms: High Dose; Low Dose
Drug: Placebo — Pharmaceutical form: Injection solution Route of administration: subcutaneous
  Arms: Placebo

SUMMARY:
This is an interventional, randomized, double blind, parallel group, placebo-controlled, Phase 2b, 3-arm study to assess the effect of pegylated-recombinant-human interleukin-2 (rezpegaldesleukin) in adult participants with severe to very severe alopecia areata.

The estimated duration includes a screening period of up to 35 days, a 36-week treatment period, an optional 16-week treatment extension period, and a 24-week follow-up period. The maximum study duration is approximately 81 weeks for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are at least 18 years and ≤60 years for males (≤70 years of age for females) old at the time of informed consent
* Diagnosis of Alopecia Areata (AA) severity at screening and baseline:

  1. severe to very severe AA (≥ 50% scalp involvement) as measured using the SALT score
  2. Documented history over 6 months with no spontaneous improvement prior to baseline
  3. Current episode of severe to very severe AA of less than 8 years
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at screening and baseline.
* While on investigational product and for at least 30 days after taking the last dose of investigational product (IP), WOCBP who engage in activity in which conception is possible must use approved highly effective contraceptive method(s). For male patient with partner that is WOCBP in which conception is possible, male patient must agree to use approved highly effective contraceptive method(s).
* Able to complete patient questionnaires
* Able and willing to comply with requested study visits and procedures
* Able and willing to provide written informed consent
* Able to communicate, read and/or understand the local language

Exclusion Criteria:

* Men and women (of reproductive potential) unwilling to use birth control and women who are pregnant or breastfeeding.
* Patient has primarily "diffuse" type AA (characterized by diffuse hair shedding).
* Presence of another form of alopecia.
* Prior use of any of the following treatments:

  1. aldesleukin
  2. investigational IL-2 analog
  3. oral Janus kinase (JAK) inhibitor for any indication, including, but not limited to, baricitinib, upadacitinib, abrocitinib, tofacitinib, and ruxolitinib, whether marketed or investigational
  4. systemic immune-modulating biologic therapy (including, but not limited to, dupilumab, tralokinumab, lebrikizumab, nemolizumab, rocatinlimab, rituximab, ocrelizumab, ofatumumab, belimumab, daxdilimab, etc.) whether marketed or investigational
* History of cancer or lymphoproliferative disease within 5 years prior to Day 1. Note: Patients with successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma with no evidence of metastatic disease for 3 years and/or localized carcinoma in situ of the cervix with no evidence of recurrence within the 3 years prior to Day 1 are not to be excluded.
* Current infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at screening.
* Other skin conditions that would interfere with study assessments of AA

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in Severity of Alopecia Tool (SALT) score at Week 36 | Baseline and Week 36
  The SALT score is the sum of percentage of hair loss in all areas with a maximum score of 100 (higher score indicates greater hair loss).

SECONDARY OUTCOMES:
Percent change from baseline in SALT score | Baseline and Weeks 12, 16, 20, 24, 28, and 32
  SALT score is the sum of percentage of hair loss in all areas with a maximum score of 100 (higher score indicates greater hair loss).
Proportion of patients achieving improvement in Severity of Alopecia Tool (SALT) ≥ 50%/75%/90% | Baseline and Weeks 12, 16, 20, 24, 28, 32, and 36
  Proportion of patients achieving improvement of ≥ 50%/75%/90% in Severity of Alopecia Tool (SALT) relative to their baseline score (SALT50/75/90). SALT score is the sum of percentage of hair loss in all areas with a maximum score of 100 (higher score indicates greater hair loss).
Proportion of patients achieving an absolute SALT score ≤ 10/20/30/50 | Baseline and Weeks 12, 16, 20, 24, 28, 32, and 36
  Proportion of patients achieving an absolute SALT score of ≤ 10/20/30/50. SALT score is the sum of percentage of hair loss in all areas (higher score indicates greater hair loss). Total percentage of patients with absolute SALT score of ≤ 10/20/30/50 will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (23):
- United States (10):
  - Nektar Investigative Site, Northridge, California
  - Nektar Investigative Site, Atlanta, Georgia
  - Nektar Investigative Site, Gurnee, Illinois
  - Nektar Investigative Site, Indianapolis, Indiana
  - Nektar Investigative Site, Clinton Township, Michigan
  - Nektar Investigative Site, Portsmouth, New Hampshire
  - Nektar Investigative Site, New York, New York
  - Nektar Investigative Site, Camp Hill, Pennsylvania
  - Nektar Investigative Site, Frisco, Texas
  - Nektar Investigative Site, Pflugerville, Texas
- Canada (5):
  - Nektar Investigative Site, Surrey, British Columbia
  - Nektar Investigative Site, Markham, Ontario
  - Nektar Investigative Site, Oakville, Ontario
  - Nektar Investigative Site, Richmond Hill, Ontario
  - Nektar Investigative Site, Sherbrooke, Quebec
- Poland (8):
  - Nektar Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Nektar Investigative Site, Nowa Sól, Lubusz Voivodeship
  - Nektar Investigative Site, Warsaw, Masovian Voivodeship
  - Nektar Investigative Site, Gdansk, Pomeranian Voivodeship
  - Nektar Investigative Site, Katowice, Silesian Voivodeship
  - Nektar Investigative Site, Sosnowiec, Silesian Voivodeship
  - Nektar Investigative Site, Olsztyn, Warmian-Masurian Voivodeship
  - Nektar Investigative Site, Szczecin, West Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: No